CLINICAL TRIAL: NCT00351286
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Oral L-Citrulline Compared to Placebo in Patients Taking Background Simvastatin 40 mg qD and With Peripheral Arterial Disease Including Intermittent Claudication
Brief Title: Efficacy Study of Oral L-Citrulline in Patients Taking Simvastatin With Peripheral Arterial Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Angiogenix (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANGX-1039-02
Record Dates: First submitted 2006-07-10; First posted 2006-07-12 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-07

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: peripheral arterial disease; peripheral vascular disease; claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases | interventions — Citrulline

INTERVENTIONS:
Drug: L-citrulline tablets, 1000 mg
Drug: Placebo tablets matching L-citrulline tablets
Drug: Background simvastatin at a stable dose of 40 mg qHS

SUMMARY:
To prove the combination of L-citrulline with simvastatin leads to greater improvement in the symptoms of peripheral arterial disease (PAD) than simvastatin alone by evaluating oral L- citrulline or placebo against simvastatin for improvement in treadmill walking distance in patients, 40-75 years of age, who have PAD with intermittent claudication.

DETAILED DESCRIPTION:
The primary objective of this study is to prove the combination of L-citrulline with simvastatin leads to greater improvement in the symptoms of PAD than simvastatin alone. This will be accomplished by evaluating efficacy of orally administered L-citrulline or placebo against background therapy with simvastatin for improvement in treadmill absolute claudication walking distance (ACWD) in patients, 40-75 years of age, who have PAD with intermittent claudication in Fontaine stage II and symptom-limited treadmill walking distance.

Secondary objectives include comparing the combination therapy to simvastatin alone for improvement in treadmill pain-free walking distance (PFWD) and ischemic window.

Other secondary objectives include evaluating the safety and tolerability of L-citrulline alone or combined with simvastatin in this patient population and assessing the effects of treatment on quality of life (QOL) as measured by two QOL instruments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 40-75 years of age
2. If female, post-menopausal for the past year, surgically sterile (i.e., tubal ligation, hysterectomy), or using an adequate method of birth control (i.e., oral contraceptives, double barrier method, IUD cover, sterilized partner, or other method deemed appropriate by Investigator)
3. If male capable of fathering children, using an adequate method of birth control (i.e., condom or partner using adequate method of birth control)
4. Peripheral arterial disease with stable, reproducible, intermittent claudication and symptom-limited treadmill walking distance of at least 6 months duration
5. Rest ankle-brachial index (ABI) ≤0.90 and 10 mm Hg decrease in ankle pressure 1 minute after completing the ETT
6. ACWD on a standardized (Skinner-Gardner protocol) ETT ≥50 m (164 feet) but ≤300 m (984 feet) determined by the average result on two consecutive ETTs performed at least 7 days apart during the screening phase (Fontaine stage II)
7. ACWD variability <25% between two consecutive ETTs performed at least 7 days apart during the screening phase. The percent variability is calculated by the difference of the two walking distances divided by the greater of the two walking distances multiplied by 100%. If the variability exceeds 25% a third ETT may be performed and the variability between the second and third test used to determine baseline and inclusion criteria
8. Willingness to receive dietary counseling and follow a low-cholesterol diet during the study
9. Ability to give written informed consent and has signed a written informed consent form approved by the Investigator's Independent Ethics Committee (IEC)

Exclusion Criteria:

1. Critical limb ischemia (defined as presence of rest pain requiring analgesics for more than 2 weeks or the presence of lower limb ulcers or gangrene)
2. Coronary artery or peripheral artery angioplasty or surgical limb arterial bypass within the last 3 months
3. Any previous amputation on the lower limbs
4. Anticipated requirement of surgical or percutaneous revascularization within 3 months of randomization
5. Currently participating in a supervised exercise regimen
6. Stroke, myocardial infarction, or deep-vein thrombosis within the last 3 months
7. Non-atherosclerotic PAD (e.g., thromboangiitis obliterans)
8. Known abdominal aortic aneurysm ≥4.5 cm
9. Unstable angina pectoris within the last 3 months
10. Congestive heart failure (New York Heart Association Class III or IV) despite treatment
11. Severe, uncontrolled hypertension (sitting systolic blood pressure >180 mm Hg or sitting diastolic blood pressure >95 mm Hg)
12. Anemia (hemoglobin <10 g/dL in women and 11 g/dL in men) or any clinically significant bleeding episode within the last year
13. Abnormal platelet count (platelets >150,000/mm3 or <60,000/mm3)
14. Type I diabetes mellitus or Type II diabetes mellitus if it is accompanied by diabetic peripheral neuropathy
15. Morbid obesity (body mass index >40 kg/m2)
16. Severe renal insufficiency (creatinine >221 µmol/L (2.5 mg/dL))
17. Severe hepatic insufficiency (ALT [SGPT] and AST [SGOT] ≥ 3x upper limit of normal on two separate tests
18. Any disorder that would affect the interpretation of ETT results
19. Use of medications that are not allowed and which cannot be discontinued during the study
20. Participation in an investigational drug or device study within previous 30 days
21. Underlying disease other than PAD resulting in a life expectancy of less than 1 year
22. If female, breast feeding, pregnancy confirmed by a positive serum pregnancy test, or using inadequate birth control
23. Other conditions that could impair informed consent or compliance

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2006-03

PRIMARY OUTCOMES:
Change in absolute claudication walking distance from baseline to end of 12-week double-blind treatment period.

SECONDARY OUTCOMES:
Change in pain-free walking distance
Changes in QOL scores from baseline to 12 and 36 weeks
Change in absolute claudication walking distance from baseline to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Spickler, MD, PhD, Study Chair — Angiogenix
Locations (10):
- Russia (10):
  - Municipal Healthcare Institution, Gatchina Central District Hospital, Gatchina, Russia
  - Russian State Medical University at Filatov City Hospital #15, Moscow, Russia
  - Vishnevsky Institute of Surgery, Russian Medical Academy of Science, Moscow, Russia
  - Municipal Prophylaxis and Treatment Institution, City Hospital #13, Nizhny Novgorod, Russia
  - St. Petersburg State Healthcare Institution, Research for Emergency Medical Care, Saint Petersburg, Russia
  - St. Petersburg State Healthcare Institution, Hospital #2, Saint Petersburg, Russia
  - St. Petersburg State Healthcare Institution, Hospital #26, Saint Petersburg, Russia
  - State Educational Institution of Higher Professional Education, Saint Petersburg, Russia
  - St. Petersburg State Healthcare Institution, Pokrovskaya Hospital, Saint Petersburg, Russia
  - Municipal Medical Institution City Hospital #1 of Saratov, Saratov, Russia